CLINICAL TRIAL: NCT00845832
Title: A Randomized, Active Controlled, Double-blind, Study to Compare the Safety and Reduction in Disease Activity With the Combination of Rituximab (MabThera®)and Tocilizumab (RoActemra®) Versus Tocilizumab in Patients With Active Rheumatoid Arthritis With an Incomplete Response to Methotrexate
Brief Title: A Study of Combination Treatment With MabThera (Rituximab) and RoActemra (Tocilizumab) Versus RoActemra in Patients With Rheumatoid Arthritis With an Incomplete Response to Methotrexate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early because of a related decision to stop the development of ocrelizumab in rheumatoid arthritis.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX21956; 2008-005525-11
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: tocilizumab [RoActemra/Actemra]
- 2 (Active Comparator)
  Interventions: Drug: Placebo; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: Placebo — iv on days 1 and 15 (Parts 1 and 2)
  Arms: 2
Drug: rituximab [MabThera/Rituxan] — 0.5g iv on days 1 and 15 (Parts 1 and 2)
  Arms: 1
Drug: tocilizumab [RoActemra/Actemra] — 2mg/kg-8mg/kg iv in Part 1 and selected dose in Part 2, on weeks 4, 8 and 12---Arm 1\n8mg/kg iv on weeks 4,8 and 12 (Parts 1 and 2)--- Arm 2

SUMMARY:
This 2 part study will investigate the safety, tolerability and efficacy of MabT hera in combination with RoActemra in patients with active rheumatoid arthritis despite a stable dose of methotrexate. In Part 1 of the study, patients will be randomized to receive either MabThera 0.5g iv or placebo on days 1 and 15, follo wed by RoActemra at one of the ascending doses between 2mg/kg and 8mg/kg at week s 4, 8 and 12 (MabThera arm) or 8mg/kg (placebo arm). In Part 2, additional pati ents will be randomized to one of 2 groups to receive MabThera 0.5g on days 1 an d 15 followed by the selected dose (from Part 1)of RoActemra at weeks 4, 8 and 1 2, or placebo on days 1 and 15 followed by RoActemra 8mg/kg at weeks 4,8 and 12.

All patients will then be eligible to receive extension treatment withRoActemra every 4 weeks. The anticipated time on study treatment is 12 months, and the tar get sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* rheumatoid arthritis, functional status I-III;
* SJC>=4 (28 joint count) and TJC>=4 (28 joint count) at screening and baseline;
* RF and/or anti-CCP positive;
* may have failed up to 1 approved anti-TNF agent (infliximab, etanercept or adalimumab);
* inadequate response to methotrexate, at a dose of 7.5-25mg weekly for at least 12 weeks, at a stable dose for past 4 weeks.

Exclusion Criteria:

* rheumatic autoimmune disease other than rheumatoid arthritis, or significant systemic involvement secondary to rheumatoid arthritis;
* history of, or current, inflammatory joint disease other than rheumatoid arthritis;
* diagnosis of juvenile idiopathic arthritis and/or rheumatoid arthritis before age 16;
* significant cardiac or pulmonary disease;
* previous treatment with any biologic agent for rheumatoid arthritis (other than infliximab, etanercept or adalimumab).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- France (4):
  - Le Kremlin-Bicêtre
  - Montpellier
  - Paris
  - Strasbourg
- Germany (4):
  - Berlin
  - Cologne
  - Heidelberg
  - Würzburg
- Greece (2):
  - Athens
  - Thessaloniki
- Netherlands (2):
  - Amsterdam
  - Leiden
- Poland (3):
  - Bytom
  - Lublin
  - Poznan
- Spain (4):
  - Santander, Cantabria
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Seville, Sevilla
- Switzerland (2):
  - Bern
  - Lausanne
- United Kingdom (2):
  - Newcastle upon Tyne
  - Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg): Participants received placebo intravenously (iv) on Days 1 and 15 followed by TCZ 8 mg/kg iv at Weeks 4, 8, 12 and 16. Participants also continued to receive a stable dose of methotrexate, between 7.5 and 25 mg/week orally or parenterally, as prescribed by the physician and in accordance with the local label. Participants also received a stable dose of folic acid.
- Rituximab (0.5 Grams [g]) + TCZ (2 mg/kg): Participants received rituximab 0.5 g iv on Days 1 and 15 followed by TCZ 2 mg/kg iv at Weeks 4, 8, 12 and 16. Participants also continued to receive a stable dose of methotrexate, between 7.5 and 25 mg/week orally or parenterally, as prescribed by the physician and in accordance with the local label. Participants also received a stable dose of folic acid.
- Rituximab (0.5 g) + TCZ (4 mg/kg): Participants received rituximab 0.5 g iv on Days 1 and 15 followed by TCZ 4 mg/kg iv at Weeks 4, 8, 12 and 16. Participants also continued to receive a stable dose of methotrexate, between 7.5 and 25 mg/week orally or parenterally, as prescribed by the physician and in accordance with the local label. Participants also received a stable dose of folic acid.
Period: Treatment Period
Arm/Group | Placebo + Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg) | Rituximab (0.5 Grams [g]) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Started | 4 | 10 | 10
Completed | 3 | 7 | 10
Not Completed | 1 | 3 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Period: Safety Follow-Up
Arm/Group | Placebo + Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg) | Rituximab (0.5 Grams [g]) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Started | 3 (One participant from this group was re-assigned to TCZ (4 mg/kg) group.) | 9 (All participants who withdrew from study were asked to return for safety follow-up.) | 12 (One participant each from the placebo and TCZ (2 mg/kg) groups were re-assigned to this group.)
Completed | 2 | 9 (One participant from this group was re-assigned to TCZ (4 mg/kg) group.) | 12
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Extended Safety Follow-Up
Arm/Group | Placebo + Tocilizumab (TCZ) 8 Milligrams Per Kilogram (mg/kg) | Rituximab (0.5 Grams [g]) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Started | 2 | 5 (Only participants who remained B cell depleted required extended safety follow-up.) | 7 (Only participants who remained B cell depleted required extended safety follow-up.)
Completed | 2 | 5 | 0
Not Completed | 0 | 0 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Safety population: All participants who were randomized and received any part of an infusion of study medication; participants who received the incorrect therapy from that intended were summarized in the group according to the therapy actually received for the majority of the time through Week 48.
Groups:
- Placebo + TCZ (8 mg/kg): Participants received placebo iv on Days 1 and 15 followed by TCZ 8 mg/kg iv at Weeks 4, 8, 12 and 16. Participants also continued to receive a stable dose of methotrexate, between 7.5 and 25 mg/week orally or parenterally, as prescribed by the physician and in accordance with the local label. Participants also received a stable dose of folic acid.
- Rituximab (0.5 g) + TCZ (2 mg/kg): Participants received rituximab 0.5 g iv on Days 1 and 15 followed by TCZ 2 mg/kg iv at Weeks 4, 8, 12 and 16. Participants also continued to receive a stable dose of methotrexate, between 7.5 and 25 mg/week orally or parenterally, as prescribed by the physician and in accordance with the local label. Participants also received a stable dose of folic acid.
- Total: Total of all reporting groups
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg) | Total
Number analyzed (Participants) | 3 | 9 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.02) | 48.2 (10.50) | 50.0 (6.97) | 48.3 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10 | 20
  Male | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) at Week 16 Assessed Using Disease Activity Score Based on 28 Joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR)
Description: The Disease Activity Score based on 28 joint count (DAS28) and Erythrocyte Sedimentation Rate (ESR), is a measure of the participant's disease activity. It is based on the Tender Joint Count (TJC [28 joints]), Swollen Joint Count (SJC [28 joints]), participant's global assessment of disease activity (PtGA) Visual Analog Scale (VAS) in millimeters (mm), and ESR in millimeters per hour (mm/hour). DAS28-ESR scores range from 0 - 10. Definition of LDA was based on DAS28-ESR scores. To achieve LDA the DAS28-ESR had to be (less than or equal to) ≤ 3.2.
  DAS28-ESR equals (=) (0.56 times (*) (square root)√ TJC plus (+) (0.28 * √ SJC + (0.70 * ln(ESR))+(0.014 * (Global Health) GH)
  Where:
  TJC = based on 28 joints SJC = based on 28 joints ESR = erythrocyte sedimentation rate in mm/hour GH = participant's global assessment of disease activity ln = natural log
Time Frame: Week 16
Population: Intent-to-Treat (ITT) Population: all randomized participants who received any part of an infusion of study medication. Last observation carried forward (LOCF) used for TJC and SJC, ESR and PtGA. If DAS28-ESR value was missing LDA was missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 4 | 9 | 10
percentage of participants | 50.0 | 11.1 | 20.0

2. Secondary Outcome: Percentage of Participants Achieving Remission at Week 16 Assessed Using DAS28-ESR
Description: The DAS28-ESR score is a measure of the participant's disease activity. It is based on the TJC (28 joints), SJC (28 joints), participant's global assessment of disease activity (mm), and ESR (mm/hour). DAS28-ESR is expressed on a unit on a scale with the minimum score=0 (best) to maximum score=10 (worst). Remission was defined as DAS28-ESR less than (<) 2.6
Time Frame: Week 16
Population: ITT Population; LOCF used for TJC, ESR, and PtGA. If the DAS28-ESR value was missing then remission or LDA was missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 4 | 9 | 10
percentage of participants | 0.0 | 0.0 | 10.0

3. Secondary Outcome: Percentage of Participants by European League Against Rheumatism (EULAR) Response Category at Week 16
Description: DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline (greater than) >1.2 with DAS28 ≤3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or DAS28-ESR >5.1 or change from baseline >0.6 to ≤1.2 with DAS28 ≤5.1; nonresponders: change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with DAS28 >5.1.
Time Frame: Week 16
Population: ITT Population; No imputation used for TJC, SJC, ESR, and PtGA. EULAR response was set to missing when the DAS28 score was missing.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 4 | 9 | 9
percentage of participants
  No Response | 0.0 | 22.2 | 11.1
  Moderate Response | 50.0 | 66.7 | 66.7
  Good Response | 50.0 | 11.1 | 22.2

4. Secondary Outcome: Change From Baseline in DAS28-ESR
Description: The DAS28-ESR score is a measure of the participant's disease activity. It is based on the TJC (28 joints), SJC (28 joints), participant's global assessment of disease activity (mm), and ESR (mm/hour). DAS28-ESR is expressed as a score on a scale with the minimum score=0 (best) to maximum score=10 (worst).
  DAS28-ESR scores were calculated as follows: DAS28-ESR = (0.56 * √TJC)+(0.28 * √SJC)+(0.70 * ln(ESR))+(0.014 * GH).
  No imputation used for tender and swollen joint counts, ESR, and patient's global assessment of disease activity VAS.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: ITT Population; number (n) = number of participants analyzed at the specified visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 4 | 10 | 10
units on a scale
  Week 4 (n=4,9,10) | -1.9 (1.73) | -0.7 (1.44) | -1.0 (0.72)
  Week 8 (n=4,10,10) | -2.7 (0.55) | -0.5 (1.33) | -1.9 (1.31)
  Week 12 (n=4,10,9) | -2.7 (0.57) | -1.2 (1.60) | -2.3 (1.36)
  Week 16 (n=4,9,9) | -3.0 (0.80) | -1.8 (1.44) | -2.3 (1.25)
  Week 20 (n=4,9,9) | -3.6 (0.70) | -2.2 (1.16) | -2.7 (1.45)
  Week 24 (n=4,9,8) | -3.5 (1.28) | -2.2 (1.14) | -2.9 (1.34)
  Week 32 (n=4,9,8) | -2.6 (1.62) | -3.1 (1.92) | -3.3 (1.83)
  Week 40 (n=3,8,8) | -2.6 (1.24) | -2.2 (1.63) | -2.7 (1.02)
  Week 48 (n=4,8,7) | -3.3 (1.84) | -2.9 (1.50) | -3.0 (1.24)

5. Secondary Outcome: Clinical Disease Activity Index Scores
Description: The Clinical Disease Activity Index (CDAI) score was calculated according to the following formula: CDAI = SJC + TJC + GH/10 + EGA/10
  Where:
  SJC = swollen joint count based on 28 joints; TJC = tender joint count based on 28 joints; GH = Participant's global assessment of disease activity; EGA = evaluator's (physician's) global assessment of disease activity. CDAI scores range from 0-76 and the following cut-off points for different disease activity states have been used: high disease activity >22; moderate disease activity >10 and ≤22; LDA >2.8 and ≤10; and remission ≤ 2.8. No imputation used for TJC, SJC, Patient's Global Assessment of Disease Activity VAS and Physicians global assessment of disease activity VAS.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 4 | 10 | 10
units on a scale
  Baseline (n=4, 10, 10) | 37.7 (4.59) | 36.4 (9.16) | 33.0 (7.69)
  Week 4 (n=4, 8, 10) | 21.2 (14.19) | 23.4 (12.38) | 20.0 (6.97)
  Week 8 (n=4,10,10) | 14.6 (4.38) | 29.4 (14.91) | 15.5 (9.96)
  Week 12 (n=4,10, 9) | 16.3 (10.52) | 23.2 (12.47) | 13.4 (8.40)
  Week 16 (n=4,10, 9) | 9.5 (5.70) | 19.5 (15.42) | 12.7 (8.32)
  Week 20 (n=4, 8, 9) | 10.8 (4.46) | 15.4 (7.76) | 11.6 (6.64)
  Week 24 (n=4, 9, 8) | 9.2 (6.71) | 12.6 (3.98) | 10.9 (5.47)
  Week 32 (n=4, 9, 8) | 15.2 (10.42) | 11.5 (13.14) | 9.3 (9.42)
  Week 40 (n=3, 8, 8) | 20.3 (8.35) | 17.9 (16.40) | 11.8 (5.31)
  Week 48 (n=4, 7, 8) | 11.6 (10.11) | 12.8 (12.15) | 7.1 (6.41)

6. Secondary Outcome: Simplified Disease Activity Index (SDAI) Scores
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), Participant and Physician assessed global disease activity (assessed on 0-100 mm VAS; higher scores = greater affection due to disease activity), and ESR (mm/hour). SDAI total score ranged from 0 to 86. Higher scores indicated greater disease activity.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, 24, 32, 40, and 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline to Week 48 in SJC and TJC
Description: An assessment of 28 joints for swelling and tenderness will be made. Joints will be assessed and classified as swollen (1)/not swollen (0) and tender(1)/not tender (0) by pressure and joint manipulation on physical examination. Joint prosthesis, arthrodesis or fused joints were not taken into consideration for swelling or tenderness. The 28 joints assessed comprise shoulders (2 joints), elbows (2 joints), wrists (2 joints), metacarpophalangeal joints on digits 1-5 (10 joints), interphalangeal on digit 1 (2 joints), proximal interphalangeal joints on digits 2-5 (8 joints), and knees (2 joints).
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline to Week 48 in Health Assessment Questionnaire (HAQ)
Description: The Stanford Health Assessment Questionnaire disability index specific for rheumatoid arthritis was completed by the participants for efficacy assessments.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline to Week 48 in C-Reactive Protein (CRP)
Description: CRP is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline to Week 48 in ESR
Description: ESR is an acute phase reactant and is a measure of inflammation.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline to Week 48 in Physician's Global Assessment of Disease Activity
Description: Physician Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity and 100 mm= maximum disease activity. The physician marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline to Week 48 in Participant's Global Assessment of Disease Activity
Description: Participant's Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no disease activity and 100 mm = maximum disease activity. The participant marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline to Week 48 in Participant's Assessment of Pain
Description: Participant's Global Assessment of Disease Activity was measured on a 0 to 100 mm VAS, with 0 mm = no pain and 100 mm = maximum pain. The participant marked the line according to their assessment and the distance from the left edge was measured.
Time Frame: Baseline and Week 48
Population: Data were not collected because the study was terminated early.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded throughout the study from the date of first study drug administration until 48 weeks of treatment period and for those in the Safety follow up population until the end of follow up period.
Description: Participants who received the incorrect therapy from that intended were summarized in the group according to the therapy actually received for the majority of the time through Week 48. 1 participant each from Placebo + TCZ (8 mg/kg) and Rituximab (0.5 g) + TCZ (2 mg/kg) groups was included in Rituximab (0.5 g) + TCZ (4 mg/kg) group.
Arm/Group | Placebo + TCZ (8 mg/kg) | Rituximab (0.5 g) + TCZ (2 mg/kg) | Rituximab (0.5 g) + TCZ (4 mg/kg)
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/9 | 3/12
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + TCZ (8 mg/kg) (N=3) | Rituximab (0.5 g) + TCZ (2 mg/kg) (N=9) | Rituximab (0.5 g) + TCZ (4 mg/kg) (N=12)
Chest pain (General disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + TCZ (8 mg/kg) (N=3) | Rituximab (0.5 g) + TCZ (2 mg/kg) (N=9) | Rituximab (0.5 g) + TCZ (4 mg/kg) (N=12)
Upper respiratory tract infection (Injury, poisoning and procedural complications) | 0 | 3 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Bronchitis (Infections and infestations) | 0 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 1 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infected bites (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 3 | 1
Asthenia (General disorders) | 0 | 1 | 2
Oedema peripheral (General disorders) | 2 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Essential tremor (Nervous system disorders) | 0 | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Corneal erosion (Eye disorders) | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1
Presbyopia (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Genital ulceration (Reproductive system and breast disorders) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 1 | 0
Asthma (Immune system disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Occipital Neuralgia (left) (Nervous system disorders) | 0 | 3 | 0
Occipital Neuralgia (right) (Nervous system disorders) | 0 | 1 | 0
Aphthous stomatitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 1 | 0
Rash (General disorders) | 0 | 1 | 0
Cervix Disorder (General disorders) | 0 | 1 | 0
Tooth Ache (General disorders) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Pyrexia (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.